CLINICAL TRIAL: NCT06146504
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of an Anti-Fungal Supplement
Brief Title: Clinical Study to Evaluate the Efficacy of an Anti-Fungal Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CanXida (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20369
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Candida Systemic; Candida Albicans Infection; Candida Infection
MeSH Terms: conditions — Candidiasis, Invasive; Candidiasis

STUDY DESIGN:
Intervention Model Description: Group A = the intervention group Group B = the placebo group
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be double-blinded in that the study participants and the Citruslabs team will be blinded to the intervention or product allocation. Only the sponsor will know which product contains the active ingredients. After the study analysis is complete, the allocation will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CanXida Supplement (Experimental): All participants will adhere to the following treatment regime:
  Day 1-7: 1 tablet per day Day 8-22: 2 tablets per day Day 23- 84: 3 tablets per day
  The product should always be taken with the first meal of the day.
  Interventions: Dietary Supplement: CanXida Remove (Formula RMV)
- Placebo (Placebo Comparator): All participants will adhere to the following treatment regime:
  Day 1-7: 1 tablet per day Day 8-22: 2 tablets per day Day 23- 84: 3 tablets per day
  The product should always be taken with the first meal of the day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CanXida Remove (Formula RMV) — Supplement composed of a 12 ingredient anti-fungal, anti-bacterial & anti-parasite formula.
  Arms: CanXida Supplement
Other: Placebo — Placebo product containing Dicalcium Phosphate, Magnesium Stearate, Stearic Acid, Croscarmellose Sodium, and Silica.
  Arms: Placebo

SUMMARY:
This is a virtual, double-blind, two-arm, randomized, placebo-controlled clinical trial that will last 12 weeks. Participants will take the CanXida Remove Candida Cleansing Formula RMV or a placebo product daily and complete questionnaires at Baseline, Week 6, and Week 12. Candida microbiome testing will be conducted via stool sample at Baseline and Week 12.

The participants will all be blinded to the name of the test brand.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-50.
2. Female.
3. Self-reported recurrent vaginal issues, including:

   * Itching and irritation in and around the vaginal area.
   * Burning sensation during urination or sexual intercourse.
   * Abnormal discharge (e.g. thicker, white, and curd-like in appearance, odorless, or with a mild yeasty smell.
   * Redness and swelling of the vulva and surrounding skin
   * Pain or discomfort in the vaginal area or lower abdomen.
   * Urinary tract infections
   * Vaginal thrush
4. May also experience issues with fatigue, lethargy, and gut or digestive issues.
5. Willing to provide two stool samples during the study.
6. Willing to adhere to the study protocol.
7. Willing to avoid introducing any products or any new forms of regular medication or supplements that target candida overgrowth, gut health, or vaginal health for the duration of the study.

Exclusion Criteria:

1. Anyone with severe chronic conditions including oncological conditions, psychiatric disease, diabetes, or other.
2. Anyone with known severe allergic reactions or is allergic to the test product or placebo ingredients.
3. Currently taking any antibiotics or will be during the trial period.
4. Anymore diagnosed with a sexually transmitted disease within the last three months e.g. Chlamydia, trichomoniasis, gonorrhea, genital herpes
5. Women who are pregnant, breastfeeding, or attempting to become pregnant.
6. Having any planned invasive medical procedures during the study period.
7. Currently participating in any other clinical study.
8. History of substance abuse.
9. Unwilling to follow the study protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Changes in growth of candida in the gut. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via gut microbiome analysis. Participants will provide a stool sample for the analysis.

SECONDARY OUTCOMES:
Changes in vaginal health symptoms. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires. Questionnaires will use a Likert scale (0-5 scale) to measure changes in vaginal itching, vaginal discharge, vaginal discomfort. On the scale, 0= the least favourable score and 5= the most favourable score.
Changes in scores on the Gastrointestinal Symptom Rating Scale (GSRS). [Timeframe: Baseline to Week 12] | 12 weeks
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Changes in scores on the Bristol Stool Scale. [Timeframe: Baseline to Week 12] | 12 weeks
  The Bristol Stool Scale is a scale that classifies stools, ranging from the hardest to the softest. Experts consider types 1 and 2 to be uncharacteristically hard and indicative of constipation, while types 6 and 7 are unusually loose and may indicate diarrhea. Medical professionals generally consider types 3, 4, and 5 to be the most typical.
Changes in self-reported energy levels. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. 0= the most favourable and 5= the least favourable response.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided